CLINICAL TRIAL: NCT06005025
Title: The Effect of Counselling and Follow-up After Breast Cancer Awareness Education on Early Diagnosis and Healthy Lifestyle Behaviours: 'Reduce Risks, Increase Life Chances'
Brief Title: Examination of the Effect of Counselling and Follow-up After Breast Cancer Awareness Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Collaborators: Mersin University (Other)
Responsible Party: Principal Investigator, Gamze BOZKUL, Principal Investigator (Research Assistant), Tarsus University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: TU-BOZKUL-003
Record Dates: First submitted 2023-08-08; First posted 2023-08-22 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer; Nurse; Education; Counselling; Follow-up
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: The study was a prospective, parallel, two-arm (1:1), randomised controlled experimental study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Firstly, the names of the personnel will be listed alphabetically. A number will be written opposite each personnel and the number of 160 personnel will be determined from the total number of administrative personnel with high risk level by randomisation generated by an independent researcher in the computer environment. The sequence number of the personnel determined by randomisation will be divided into group A (study) and group B (control) in the computer environment and the information showing that they are assigned to group A and B according to the randomisation table will be placed in an opaque envelope. This envelope will be kept by the coordinator researcher and when the staff is approached for training, it will be learnt which group the staff is in. Since all personnel will be trained, the personnel will be blinded. The data will be computerised by the researcher and a biostatistician independent of the research will blind the groups unknowingly
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REMİNDER MESSAGE (Experimental): All participants will be given one-hour training on breast cancer, modifiable and non-modifiable risk factors for breast cancer, symptoms of breast cancer, screening programmes and breast self-examination. In addition to the presentation, breast self-examination will be applied one-to-one with a breast examination model. This group will be counselled for 6 months after the training and a reminder message will be sent via SMS on Monday every week as "Check your modifiable risk factors for breast cancer" and their feedback will be received.
  Interventions: Other: Reminder message
- CONTROL GROUP (No Intervention): All participants will be given one-hour training on breast cancer, modifiable and non-modifiable risk factors for breast cancer, symptoms of breast cancer, screening programmes and breast self-examination. In addition to the presentation, breast self-examination will be applied one-to-one with a breast examination model. There will be no additional practice outside the training.

INTERVENTIONS:
Other: Reminder message — Experimental group will be counselled for 6 months after the training and a reminder message will be sent via SMS on Monday every week as "Check your modifiable risk factors for breast cancer" and their feedback will be received.
  Arms: REMİNDER MESSAGE

SUMMARY:
The aim of the study was to examine the effect of counselling and follow-up after education on the risks and prevention methods of breast cancer on early diagnosis behaviours and healthy lifestyle behaviours. The population of the study will consist of female administrative staff working at Mersin University. The sample of the study will consist of 160 people. A total of 160 personnel determined by randomisation will be divided into group A (study) and group B (control) formed by the independent researcher in the computer environment. All participants will be given a one-hour training on breast cancer and will be practised with a model as well as a presentation. Group A will be counselled for 6 months after the training and a reminder message will be sent via SMS on Monday every week as "Check your modifiable risk factors for breast cancer" and their feedback will be received. In group B, no additional application will be made except for the training. The data of the study will be collected before and 6 months after the training by using the Descriptive Characteristics Form, Breast Cancer Early Diagnosis Behaviours Form, Counselling Form and Healthy Lifestyle Behaviours Scale II. The data obtained from the study will be analysed in a computer environment. Number, percentage, mean and standard deviation will be used as descriptive statistics in the evaluation of the data.

DETAILED DESCRIPTION:
The study was a prospective, parallel, two-arm (1:1), randomised controlled experimental study. The aim of the study was to examine the effect of counselling and follow-up after education on the risks and prevention methods of breast cancer on early diagnosis behaviours and healthy lifestyle behaviours. The population of the study will consist of female administrative staff working at Mersin University. The sample of the study will consist of 160 people with an effect size of 0.23, 80% power maximum 5% type 1 error and drop out rate of 10%. The sample determined by randomisation A total of 160 personnel in the group will be divided into group A (study) and group B (control) formed by the independent researcher in the computer environment. All participants will be given one-hour training on breast cancer, modifiable and non-modifiable risk factors for breast cancer, symptoms of breast cancer, screening programmes and breast self-examination. Group A will be counselled for 6 months after the training and a reminder message will be sent via SMS on Monday every week as "Check your Changeable Risk Factors for Breast Cancer" and their feedback will be received. In group B, no additional application will be made except for the training. The data of the study will be collected before and 6 months after the training by using the Descriptive Characteristics Form, Breast Cancer Early Diagnosis Behaviours Form, Counselling Form and Healthy Lifestyle Behaviours Scale II. The data obtained from the study will be analysed in a computer environment. Number, percentage, mean and standard deviation will be used as descriptive statistics in the evaluation of the data.

ELIGIBILITY:
Inclusion Criteria:

* 35 years and older,
* No visual impairment and no physical problems that would prevent breast self-examination,
* Not previously diagnosed with breast cancer,
* Accepted to participate in the research,
* Female administrative staff working at Mersin University

Exclusion Criteria:

* 35 and under,
* Visually impaired and have a physical problem that would prevent them from performing breast self-examination,
* Previously diagnosed with breast cancer,
* Willing did not agree to participate in the research,
* Female administrative staff not working at Mersin University

Min Age: 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Behaviours for Early Diagnosis of Breast Cancer | 6 months
  Breast Cancer Early Diagnosis Behaviours Form: It is a form consisting of 5 questions about the frequency of early diagnosis behaviours such as breast self-examination, clinical breast examination and mammography.
Counselling | 6 months
  Counselling Form: This is a 5-question form that includes information on the subject consulted, the number of consultations, what was recommended in the consultation, the status of referral to a health institution after the consultation and what the outcome was if referred to a health institution.
Healthy Lifestyle Behaviours | 6 months
  Healthy Lifestyle Behaviours Scale II; The scale consists of six subscales under the titles of 'health responsibility', 'physical activity', 'nutrition', 'spiritual development', 'interpersonal relationships' and 'stress management'. The higher score obtained from the scale indicates more appropriate lifestyle behaviour.

CONTACTS AND LOCATIONS:
Overall Officials: Seher Gürdil Yılmaz, Lecturer Dr., Principal Investigator — Mersin University; Gamze Bozkul, Res. Ass, Principal Investigator — Tarsus University; Gülay Altun Uğraş, Assoc.Dr., Study Director — Mersin University
Locations (1):
- Gamze Bozkul, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guo W, Fensom GK, Reeves GK, Key TJ. Physical activity and breast cancer risk: results from the UK Biobank prospective cohort. Br J Cancer. 2020 Mar;122(5):726-732. doi: 10.1038/s41416-019-0700-6. Epub 2020 Jan 10. PMID 31919405
- [Background] Gui Y, Pan Q, Chen X, Xu S, Luo X, Chen L. The association between obesity related adipokines and risk of breast cancer: a meta-analysis. Oncotarget. 2017 May 13;8(43):75389-75399. doi: 10.18632/oncotarget.17853. eCollection 2017 Sep 26. PMID 29088874
- [Background] Niehoff NM, Nichols HB, Zhao S, White AJ, Sandler DP. Adult Physical Activity and Breast Cancer Risk in Women with a Family History of Breast Cancer. Cancer Epidemiol Biomarkers Prev. 2019 Jan;28(1):51-58. doi: 10.1158/1055-9965.EPI-18-0674. Epub 2018 Oct 17. PMID 30333218
- [Background] De Cicco P, Catani MV, Gasperi V, Sibilano M, Quaglietta M, Savini I. Nutrition and Breast Cancer: A Literature Review on Prevention, Treatment and Recurrence. Nutrients. 2019 Jul 3;11(7):1514. doi: 10.3390/nu11071514. PMID 31277273
- [Background] Skouroliakou M, Grosomanidis D, Massara P, Kostara C, Papandreou P, Ntountaniotis D, Xepapadakis G. Serum antioxidant capacity, biochemical profile and body composition of breast cancer survivors in a randomized Mediterranean dietary intervention study. Eur J Nutr. 2018 Sep;57(6):2133-2145. doi: 10.1007/s00394-017-1489-9. Epub 2017 Jun 20. PMID 28634625
- [Background] Walker SN, Sechrist KR, Pender NJ. The Health-Promoting Lifestyle Profile: development and psychometric characteristics. Nurs Res. 1987 Mar-Apr;36(2):76-81. PMID 3644262
- [Background] Sonkaya Z.İ, Günay O. The impact of education given to obese and preobese university students according to the health promotion model on nutrition and physical activities. Cukurova Medical Journal. 2020;45(3):795-806.
- [Background] Global Cancer Observatory. https://gco.iarc.fr/today/data/factsheets/populations/900-world-fact-sheets.pdf , Erişim
- [Background] Promoting Cancer Early Diagnosis. https://www.who.int/activities/promoting-cancer-early-diagnosis
- [Background] Dell, D. (2020). Breast disorders. In: M.M. Harding, J. Kwong, D. Roberts, D. Hagler, C. Reinisch (Eds.) Lewis's Medical Surcigal Nursing Assesment and Management of Clinical Problems. (11th ed). St. Louis Missouri: Elsevier;1190-1211.
- [Background] Ozmen V. Breast Cancer in Turkey: Clinical and Histopathological Characteristics (Analysis of 13.240 Patients). J Breast Health. 2014 Apr 1;10(2):98-105. doi: 10.5152/tjbh.2014.1988. eCollection 2014 Apr. PMID 28331652